CLINICAL TRIAL: NCT06699498
Title: Phase II Clinical Study of Neoadjuvant Therapy With Benmelstobart Combined With Anlotinib and Chemotherapy for Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Neoadjuvant Therapy of Targeted Immunotherapy Combined With Chemotherapy for Locally Advanced HNSCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-421
Record Dates: First submitted 2024-06-16; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Neoadjuvant Therapy; PD-L1; Anlotinib
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — anlotinib; Cisplatin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): The treatment group received neoadjuvant therapy with benmelstobart, anlotinib, cisplatin, and albumin-bound paclitaxel for a total of 3 cycles.
  Surgery was performed within 2 weeks after completing neoadjuvant therapy. Adjuvant therapy was initiated within 6 weeks after surgery.
  Interventions: Drug: Benmelstobart; Drug: Anlotinib; Drug: Cisplatin; Drug: Paclitaxel for Injection （Albumin Bound）

INTERVENTIONS:
Drug: Benmelstobart — 1200mg, D1, IV,q3w
  Other Names: TQB2450
Drug: Anlotinib — 10mg，D1-14，po，q3w
Drug: Cisplatin — 60mg/m2， D1， IV，q3w
Drug: Paclitaxel for Injection （Albumin Bound） — 260mg/m2，IVgtt ，D1，q3w
  Other Names: Albumin Bound-Paclitaxel

SUMMARY:
Exploring the safety and effectiveness of neoadjuvant therapy using benmelstobart combined with anlotinib and chemotherapy for locally advanced squamous cell carcinoma of the head and neck patients.

DETAILED DESCRIPTION:
This is a single-center, Phase II study designed to treat patients with stage III/IVa head and neck squamous cell carcinoma who meet the inclusion and exclusion criteria. The neoadjuvant therapy involves the administration of benmelstobart combined with anlotinib and chemotherapy for three cycles (21 days per cycle). Surgical resection will be performed within 2 weeks after the completion of neoadjuvant therapy. Tumor tissue samples and blood samples will be collected post-surgery for ctDNA detection. If the post-surgical ctDNA test result is positive, the patient will receive standard adjuvant therapy combined with benmelstobart, along with benmelstobart maintenance therapy. If the result is negative, the patient will receive standard adjuvant therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old;
* ECOG PS score of 0-1;
* Pathologically confirmed, untreated patients with head and neck squamous cell carcinoma, classified as stage III, IVa according to AJCC (8th edition), including hypopharyngeal cancer, laryngeal cancer, and oral cancer;
* Women of childbearing age must have taken reliable contraceptive measures or undergone a pregnancy test (serum or urine) within 7 days before enrollment, with a negative result, and are willing to use appropriate contraceptive methods during the trial and for 8 weeks after the last administration of the trial drug, or have undergone sterilization. For male participants, they must agree to use appropriate contraceptive methods during the trial and for 8 weeks after the last administration of the trial drug, or have undergone surgical sterilization;
* Signed the informed consent form with their own consent and have good compliance.

Exclusion Criteria:

* Received previous PD-1/PD-L1/CTLA-4 antibody therapy;
* Tumor invasion of major blood vessels;
* Patients requiring systemic use of glucocorticoids (>10mg daily prednisone equivalent) or other immunosuppressive drugs within 14 days before administration or during treatment. Inhaled or local use of steroids and adrenal corticosteroids at doses >10mg/day prednisone equivalent are allowed in the absence of active autoimmune diseases. Adrenal corticosteroid replacement therapy not exceeding 10mg/day prednisone equivalent is also allowed;
* Presence of any history of active immune or autoimmune diseases, or known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* Active or uncontrolled severe infection (≥NCI CTCAE v5.0 Grade 2 infection) within 4 weeks before enrollment;
* Abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), tendency to bleed, or receiving thrombolytic or anticoagulant therapy; Note: Small doses of heparin (adult daily dose of 6,000-12,000 U) or small doses of aspirin (daily dose ≤ 100 mg) for preventive purposes are allowed provided that the international normalized ratio of prothrombin time (INR) is ≤ 1.5;
* Patients with imaging showing tumor invasion of vital perivascular tissue or whose tumor is likely to invade vital blood vessels during subsequent study and cause fatal bleeding as judged by the investigator;
* Patients with any signs or history of bleeding diathesis, regardless of severity;
* patients with any bleeding or hemorrhage event ≥ CTCAE Grade 2 within 4 weeks before enrollment, presence of unhealed wounds, ulcers, or fractures;

Abnormalities in major organ functions:

* Abnormal blood routine examination (received blood transfusion or blood products, or used G-CSF and other hematopoietic growth factors for correction within 14 days):

  1. Hemoglobin (HB) < 90g/L;
  2. Absolute neutrophil count (ANC) < 1.5 × 109/L;
  3. Platelets (PLT) < 100 × 109/L;

     * Abnormal biochemical examination:

  <!-- -->

  1. Total bilirubin (TBIL) > 1.5 * upper limit of normal (ULN);
  2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 × ULN;
  3. Serum creatinine (Cr) > 1.5 × ULN or creatinine clearance rate (CCr) < 60ml/min; ③ Abnormal Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) < normal lower limit (60%);

     * Abnormal thyroid function: TSH > upper limit of normal (ULN) with abnormal T3 and T4 levels;

       * Renal insufficiency: Urine routine test indicating urine protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0g;
       * Grade I or higher myocardial ischemia or myocardial infarction, arrhythmia (including QTc ≥ 480ms), and ≥ Grade 2 congestive heart failure (New York Heart Association (NYHA) classification) within 6 months before enrollment;
       * Diagnosed with other malignancies within 3 years before enrollment;
       * Patients with any severe and/or uncontrolled diseases, including:

  <!-- -->

  1. Patients with uncontrolled blood pressure (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg); Grade I or higher myocardial ischemia or myocardial infarction, arrhythmia (including QT interval ≥ 430ms), and Grade I cardiac insufficiency (NYHA classification);
  2. Active or uncontrolled severe infections;
  3. Diseases such as cirrhosis, decompensated liver disease, active hepatitis HBV or HCV;
  4. Poorly controlled diabetes (fasting blood glucose (FBG) > 10mmol/L);
  5. Urine routine test indicating urine protein ≥ 2+, and confirmed 24-hour urine protein > 1.0g;

     - Presence of long-term unhealed wounds or fractures;

     - Pulmonary hemorrhage graded > 1 by NCI CTC AE V4.0 within 4 weeks before enrollment; hemorrhage in other locations graded > 2 by NCI CTC AE V4.0 within 4 weeks before enrollment; patients with a tendency to bleed (such as active peptic ulcer) or receiving thrombolytic or anticoagulant therapy such as warfarin, heparin, or similar drugs;

     - History of gastrointestinal perforation and/or fistula within 6 months before selected treatment; or history of arterial/venous thrombotic events such as cerebrovascular accidents (including transient ischemic attacks), deep venous thrombosis, and pulmonary embolism;

     - Imaging showing tumor invasion of vital blood vessels or patients whose tumor is likely to invade vital blood vessels and cause fatal bleeding during subsequent study as judged by the investigator;

     - Clinically significant ascites, including any ascites detectable by physical examination, ascites that has been treated or still requires treatment, and patients with only a small amount of ascites shown by imaging but asymptomatic are eligible;

     - Uncontrolled metabolic disorders or other non-malignant tumor organ or systemic diseases or secondary reactions to cancer that can lead to high medical risks and/or uncertainty in survival evaluation;

     - Participated in other anti-cancer drug clinical trials within 4 weeks before enrollment;
     * Patients with a history of psychotropic drug abuse who cannot quit or have mental disorders;
     * Any accompanying diseases or other conditions that the investigator judges as seriously endangering the safety of the patient, potentially confusing the study results, or affecting the patient's completion of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-03 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Major pathological response，MPR | up to 9 weeks
  It is defined as pathological examination shows that the tissue sample has ≤10% viable tumor, i.e. the area of residual viable tumor cell region/surface area of tumor bed ≤10%.

SECONDARY OUTCOMES:
Objective response rate (ORR) evaluated by RECIST 1.1 | up to 9 weeks
  The proportion of patients whose tumors have shrunk to a certain extent and maintained for a certain period of time, including cases of complete response (CR) and partial response (PR). The tumor's objective response is assessed using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1 criteria).
Pathological complete remission rate (pCR) | up to 9 weeks
  Defined as pathological examination showing 0% viable tumor tissue (0% RVT); calculate the proportion of subjects achieving pathological complete remission (pCR).
Disease-free survival rate at 2 years | from enrollment to the end of the second year
  The proportion of subjects who experienced disease recurrence or died (from any cause) from enrollment to the end of the first year, out of the total number of subjects.
Locoregional recurrence-free survival rate (LRFS) at 2 years | from enrollment to the end of the second year
  The proportion of subjects who did not experience local or regional lymph node recurrence or death from enrollment to the end of the second year, out of the total number of subjects.
Distant metastasis-free survival rate (DMFS) at 2 years | from enrollment to the end of the second year
  The proportion of subjects who did not experience distant metastasis from enrollment to the end of the second year, out of the total number of subjects.
Overall survival rate (OS) at 2 years | from enrollment to the end of the second year
  The proportion of subjects who died from any cause from enrollment to the end of the second year, out of the total number of subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No